CLINICAL TRIAL: NCT03492008
Title: Comparison of Three Techniques of Nasogastric Tube Insertion Without Instrumentation in Anesthetised Intubated Patients: A Prospective Randomized Controlled Trial
Brief Title: Comparison of Three Techniques of Nasogastric Tube Insertion Without Instrumentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201510-1718
Record Dates: First submitted 2018-04-02; First posted 2018-04-09 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: General Anesthesia
Keywords: nasogastric tube; general anesthesia; head position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (3):
- Conventional technique (Active Comparator): Nasogastric tube
  Interventions: Other: Conventional technique
- Contralateral cricothyroid pressure (Experimental): Nasogastric tube
  Interventions: Other: Contralateral cricothyroid pressure
- Ipsilateral head turning (Experimental): Nasogastric tube
  Interventions: Other: Ipsilateral head turning

INTERVENTIONS:
Other: Conventional technique — Nasogastric tube insertion with patient's head in neutral position
  Arms: Conventional technique
Other: Contralateral cricothyroid pressure — Cricothyroid pressure is applied externally in the contralateral direction of selected nostril before nasogastric insertion.
  Arms: Contralateral cricothyroid pressure
Other: Ipsilateral head turning — Patient's head is turned to the ipsilateral side of the selected nostril before nasogastric tube insertion.
  Arms: Ipsilateral head turning

SUMMARY:
This study compares two modified techniques(contralateral cricothyroid pressure and ipsilateral head turning technique) of nasogastric tube insertion in anesthetized and intubated patients with the conventional technique.

DETAILED DESCRIPTION:
The insertion of nasogastric tube in anesthetized, paralysed and intubated unconscious patients may be difficult, with a reported failure rate of nearly 50% on the first attempt, with the head in neutral position there are many different maneuvers to facilitate the insertion of nasogastric tube published.

Our hypothesis is that contralateral cricothyroid pressure to the selected nostril for nasogastric tube insertion will be able to avoid the difficulty.

Therefore we are going to compare this technique with the conventional technique (head in neutral position) with lateral head turning group and contralateral cricothyroid pressure group We hope that the contralateral cricothyroid pressure will increase the success rate, as this will be helpful in intubated patients with neck pathology.

ELIGIBILITY:
Inclusion Criteria:

* patient who is scheduled for elective surgery under general anaesthesia requiring NGT insertion
* aged 20 to 70 years old
* with normal airway (Commack Lehane 1 or 2) and neck movements.

Exclusion Criteria:

* Patient who has nasal stenosis, nasal septal deviation, upper airway deformity, base of skull fracture, oesophageal disorders, coagulopathy, and pregnant.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Overall success rate | At induction of general anesthesia
  Percentage

SECONDARY OUTCOMES:
First attempt success rate | At induction of general anesthesia
  Percentage
Time taken to successful nasogastric tube placement | At induction of general anesthesia
  Procedure start time is defined as the time when the nasogastric tube is inserted through the nostril. The procedure end time is defined as the time of successful insertion and confirmed NGT placement or the time after two failed attempts. The outcome is measured in second.

CONTACTS AND LOCATIONS:
Overall Officials: Sook Hui Chaw, M.Med, Principal Investigator — University of Malaya

IPD SHARING:
Plan to Share IPD: No